CLINICAL TRIAL: NCT00119990
Title: Changes in Cardiovascular Hemodynamics During Peritoneal Dialysis; the Effect of Different Dialysates
Brief Title: Changes in Cardiovascular Hemodynamics During Peritoneal Dialysis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Per Ivarsen, MD, PhD, Departement of Renal Medicine, Aarhus Universityhospital, Skejb
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AA20050009
Record Dates: First submitted 2005-07-05; First posted 2005-07-14 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-12

CONDITIONS: Peritoneal Dialysis
Keywords: vasopressin; icodextrin; cardiac output
MeSH Terms: conditions — Diabetes Insipidus | interventions — Icodextrin; Dialysis Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Icodextrin (dialysate) — 2 liter of extraneal are given with one fill for 4 hours.
Drug: Physioneal (dialysate) 1.36% and 2.27% — 2 liter of Physioneal of 1.36% or 3.86% are given with one fill for 4 hours one two different days.

SUMMARY:
During peritoneal dialysis, water is removed from the body. This sometimes occurs at rates of up to 500 ml/h. During shifts with dialysate with high glucose content, an increase in blood pressure has been described. The effect upon central hemodynamics is unknown. The researchers are investigating the effects of low and high glucose dialysate and icodextrin on cardiac output, stroke volume, pulse rate and blood pressure. The researchers have hypothesized that the effects seen are induced by vasopressin.

ELIGIBILITY:
Inclusion Criteria:

* Peritoneal dialysis patients

Exclusion Criteria:

* Insulin dependent diabetes mellitus
* AV-fistula, cardial arrhythmia persistence, or severe cardiac and lung disease
* Recent infectious disease
* Severe psychiatric disease
* Hypersensitivity to icodextrin

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Changes in cardiac hemodynamics. (Cardiac Output, stroke volume, pulse rate, blood pressure and total peripheral resistance) | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Per Ivarsen, Principal Investigator — Department of Renal Medicine C, Skejby Hospital, Denmark
Locations (1):
- Deparment of Renal Medicine, Skejby Hospital, Aarhus, Denmark

REFERENCES:
- [Background] Boon D, Bos WJ, van Montfrans GA, Krediet RT. Acute effects of peritoneal dialysis on hemodynamics. Perit Dial Int. 2001 Mar-Apr;21(2):166-71. PMID 11330561